CLINICAL TRIAL: NCT04947111
Title: Serological Study of Dengue and Characterization of Immune Response in Ten Endemic and Non-Endemic Cities in Mexico
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mexican Society of Public Health (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1
Record Dates: First submitted 2021-06-26; First posted 2021-07-01 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Dengue
Keywords: Dengue Vaccines; Serologic Test
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Intervention Model Description: * Estimate the specific serotype prevalence for DENGUE Virus in groups from 5 to 35 years old in areas of low and high dengue endemicity.
  * Determine the general prevalence of antibodies (IgG) against DENGUE Virus in groups aged 5 to 35 years in areas of high and low incidence of dengue.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serological survey (Other): A blood sample will be taken to estimate the specific serotype prevalence for dengue virus in groups of 5 to 35 years in areas of low and high dengue endemicity.
  Interventions: Diagnostic Test: Estimate the distribution of antibodies by serotype by Dengue virus in areas of low and high incidence of dengue

INTERVENTIONS:
Diagnostic Test: Estimate the distribution of antibodies by serotype by Dengue virus in areas of low and high incidence of dengue — Indirect IgG ELISA to estimate seroprevalence: The seropositivity will be evaluated with the Indirect IgG ELISA following the instructions of the Panbio E-DEN 01 G manufacturer, which has a specificity of 98% and a sensitivity of 100%. In brief, 10 microliters of participant serum will be used for each assay. Each kit provides a positive and negative control, as well as three calibrators, with the respective values for quality control. Samples will be classified as positive, negative or indeterminate according to the cut-off point for each ELISA kit.
  Neutralizing antibody titers serotype-specific: To establish the type of humoral immunity that the selected city presents, the measurement of the neutralizing antibody titers will be carried out by means of the neutralization test by reducing the number of lytic plaques to 50% (PRNT50%) , using Vero cells and the following reference strains for each serotype: DENV-1 (HAWAI), DENV-2 (NEW GUINEA), DENV-3 (H-887) and DENV-4 (H-24)
  Other Names: Indirect IgG ELISA to estimate seroprevalence; PRNT to describe Serotype-specific neutralizing antibody titer

SUMMARY:
Background: Dengue continues to be a high priority disease for public health in tropical and subtropical countries, where vector control measures have not had the expected impact on transmission. The development of new vaccines opens the possibility of having an additional measure capable of preventing the development of the disease and avoiding its complications. Currently, in two of the Dengue virus (DENV) vaccines a differential behaviour of the immune response has been observed between seropositive and seronegative individuals, which makes the generation of evidence from prevalence studies in places of high and low endemicity more relevant. Objective: To determine the predominant type of humoral immune response in high areas and to estimate the serotype-specific prevalence for DENV in people groups aged 5 to 35 years living in Mexican cities with low and high dengue endemicity. Methodology: Descriptive cross-sectional study with subgroup analysis (by endemic and non-endemic areas, by age groups and by sex). Expected results: In areas of low dengue endemicity the humoral immune response against dengue is predominantly monotypic (against one serotype) while in areas of high dengue endemicity it is predominantly multitype (against two or more serotypes).

DETAILED DESCRIPTION:
Dengue is a disease of epidemiological importance in tropical and subtropical countries. The region of the Americas is one of the most affected worldwide, where nearly 500 million people are at risk of acquiring the disease from one of the four Dengue virus serotypes (DENV-1, DENV-2, DENV-3 and DENV-4) transmitted mainly by the bite of the mosquito Aedes aegypty. It is a disease subject to epidemiological surveillance based on the operational definition of a probable case of non-severe dengue, a probable case of dengue with warning signs, and a probable case of severe dengue. The clinical diagnosis is made during the febrile phase up to five days of evolution, through RT-qPCR and in the convalescence phase, six to fourteen days after the date of onset of symptoms, with an Enzyme-linked immunosorbent assay (ELISA) IgM or IgG. Although epidemiological surveillance systems are essential tools for disease description and decision-making, it has been considered that they could provide underestimated information on the burden of the disease.

About 75% of DENV infections are mild or asymptomatic, and the most common clinical manifestations are fever, headache, retro-orbital pain, myalgia, arthralgia, and nausea. Primary infection can produce a lifelong serotype-specific immune response and a cross-response against the different DENV serotypes for a period of between six months and one year (short-lived heterologous immunity), but after this time the resulting protective profile is known as a monotypic response, then, the neutralizing activity is only against one serotype. The second infection, usually caused by a different serotype, might be associated with an increased risk of developing serious manifestations; those that resolve the infection develop an antibody profile similar to that generated in the first infection (antigenic original sin), but unlike the first infection, the resulting heterologous crossed humoral immune response lasts longer; Later infections, normally asymptomatic, if carried out, intensify this profile of antibodies as a multitype response or against two or more serotypes. Although protective immunity against the Dengue virus is still being studied, it is considered that the multitype profile, developed by exposure to multiple serotypes of the virus, is the one that is related to protection against the disease and therefore it is desirable to develop by a vaccine candidate.

Another relevant aspect of dengue transmission is that the localities that develop a hyperendemic state are those where multitypic profiles should be found more frequently since these can only be generated by the circulation of more of a serotype. On the other hand, communities with the circulation of one serotype or where the circulation of more than one serotype is widely separated in time would have monotypic profiles that distinguish non-endemic communities.

Preventive measures mainly include those related to health promotion and vector control. One vaccine has been registered (CYD-TDV, yellow fever chimera 17D-DENV) and another five are under study. The World Health Organization has called for serological surveys to be carried out as key instruments to inform public policy about the prevalence of the disease and guide decision-making. This is more relevant since the CYD-TDV vaccine and TAK-003 vaccine (DENV-DENV chimera) showed a differentiated behaviour between seronegative and seropositive subjects and the CYD-TDV vaccine has been registered for exclusive use for endemic regions and localities. Additionally, an association has been reported between the vaccination history and the severity of the disease in the population under 9 years of age. Therefore, it is important to know the humoral immune response in this age group. Serological surveys have facilitated the documentation of the role of clinical, social and environmental factors in the prevalence of the disease and its heterogeneity worldwide. The prevalence of dengue in endemic areas has been reported to be around 80% while in non-endemic areas it is less than 30%. Age has also has been described as a factor associated with the prevalence of dengue in Mexico, it has been reported a prevalence of 35.7% in the group of 5-9 years, followed by 52.2% in the group of 10 to 14 years, 58.9% in the 15 to 19-year-old group, 74.1% in the 20 to 24-year-old group, 80% in the 25 to 29-year-old group and over 90% in the 30-year-old group. Infrastructure and social factors have also been documented as determinants of dengue endemicity.

Dengue seroprevalence studies carried out in Mexico have been observational studies in endemic populations; There is only one national cluster-randomized study that provides a global description of seroprevalence in endemic and non-endemic regions, and the serotype-specific neutralizing humoral response was not evaluated by Amaya-Larios et al, 2014; therefore, there is a lack of knowledge of the type of humoral immune response that occurs in endemic and non-endemic localities. Knowledge of the general characteristics of cities with monotypic or multitypic profiles will allow us to offer crucial information at various levels. For pharmaceutical companies, knowing the immune status of the country's cities will allow establishing the best places where clinical studies can be carried out to establish the efficacy and safety of vaccine candidates; For the institutions in charge of elaborating the possible public vaccination policies, knowing the general characteristics of the localities where the immune response profile and the incidence of the disease are known, will allow extrapolating this information in localities where only the incidence is known; For the international scientific community, the results of the proposed project will contribute to the knowledge of the population characteristics of the endemic transmission of dengue and its relationship with the endemic-epidemic cycles that are distinctive of the behaviour of this disease.

Research question: What is the distribution and characterization of the humoral immune response by DENV serotype in areas of low and high dengue endemicity in Mexico? Hypothesis: In areas with low dengue endemicity, the humoral response against dengue is predominantly monotypic, whereas in areas of high endemicity for dengue it is predominantly multitypic.

Objectives GENERAL

● Characterize the predominant type of humoral immune response in people 5 to 35 years of age who live in Mexican cities with low and high dengue endemicity.

SPECIFIC

* Estimate the general prevalence of antibodies (IgG) against DENV in the study population.
* Determine the neutralizing antibody titer against DENV-1, DENV-2, DENV-3 and DENV-4 in the study population.
* Determine the frequency of the type of monotypic and multitypic humoral response in cities based on their endemicity.

Methodology Study design: Descriptive cross-sectional observational study with prospective data collection.

Target population: Resident population of endemic and non-endemic urban areas for dengue.

Study population: Subjects aged 5 to 35 years resident of selected localities with high and low endemicity for dengue.

Inclusion and exclusion criteria: described below as eligibility

Sample Size Calculation: it was carried out in the OpenEpi program, Version 3 considering the prevalences reported by previous studies and extrapolating the information available from some cities on the degree of dengue endemicity for those localities in which there was no available information ( 16, 20-21) The formula for the sample size calculation was:

n = [DEFF * Np (1-p)] / [(d2 / Z21-α / 2 * (N-1) + p * (1-p)] In total, 2,421 people will need to be sampled. The selection of participants will be carried out by a two-stage sampling (by clusters of two stages) for each of the study locations. In the first stage, blocks (n = 50) will be randomly selected in each locality and later, in the second stage, a home will be selected within each block, starting with the first house on the northeast corner of the block, if this house does not accept, the community worker will continue to the right until at least one person from a household, who meets the selection criteria, agrees to participate.

Indirect IgG ELISA to estimate seroprevalence: The seropositivity will be evaluated with Indirect IgG ELISA following the instructions of the Panbio E-DEN 01 G manufacturer, which has a specificity of 98% and a sensitivity of 100%.

Neutralizing antibody titers serotype-specific: To establish the type of humoral immunity that the selected city presents, the measurement of the neutralizing antibody titers will be carried out through the neutralization test by reducing the number of lytic plaques to 50% (PRNT50%), using Vero cells and the following reference strains for each serotype: DENV-1 (HAWAI), DENV-2 (NEW GUINEA), DENV-3 (H-887) and DENV-4 (H-24).

The type of humoral immunity will be classified into monotypic immune response if only antibodies against a single DENV serotype are detected, and multitypic immune response, if antibodies are detected against more than one single DENV serotype.

Information collection and management: The information will be collected in a standard format. The survey will be filled out by the interviewer (project staff) based on the filling instructions. The information will be captured on printed surveys and managed by trained data loggers in the electronic database designed for this purpose.

The results of the laboratory tests will be managed only with the folio assigned to each participant and the results will be entered in a database made in Excel® by the laboratory staff. The database will include folio, result date and the result. The nominal information of the survey will be kept separate from the rest of the information, identifying individuals only by their folio number and protecting their identity.

The qualitative variables will be described with absolute and relative frequencies, and the quantitative variables will be described with measures of central tendency and dispersion considering the distribution of each variable. The prevalence of IgG against DENV will be determined with the respective 95% confidence intervals (95% CI) for the total study population, as well as for each locality, by age group and by sex. Similarly, the prevalence of neutralizing antibodies for specific serotypes, and the frequency of monotypic and multipic responses in these same subgroups will be determined.

Ethical considerations: This study is an investigation with minimal risk, in which only subjects who agree to participate voluntarily will be considered. For subjects of legal age, they will be asked to sign the informed consent, in which their voluntary participation is accredited; In the case of minors, the signature of the informed consent of the parent or guardian will be requested and if the minor is between 7 years and 17 years old, the signature of the informed assent will be requested.

The data security process will consist of separating the nominal information of the survey from the rest of the information, this will be stored in two tables that will be identified with a common identification key, to protect the identity of the people.

Biosafety considerations: The management of infectious biological hazardous waste is specified in this document. In general, materials in contact with viruses or blood or their derivatives will be chlorinated for 30 minutes with a 5% sodium hypochlorite solution and later they will be discarded in a red bag. The needles will be stored in a sharps container that complies with local guidelines NOM-087.

ELIGIBILITY:
Inclusion criteria:

* Subjects from 5 years to 35 years who live in the selected localities.
* Informed consent for adults or for the parents of minors who participate in the study.
* Informed assent for children and adolescents between 7 years and 17 years.

Exclusion criteria:

* Diseases that prevent consent from themselves.
* Insufficient blood sample volume to perform laboratory tests.

Ages: 5 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1960 (Estimated)
Dates: Start 2022-04-30 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with Dengue IgG antibodies | four months
  Using ELISA for IgG-Indirect, results might be positive, negative or undetermined
Ratio of neutralizing antibodies against DENV1, DENV2, DENV3 and/or DENV4 | Six months
  Using PRNT, values might be 1:20, 1:40, 1:80, 1:160, 1:320 and 1:640.
Percentage of participants with monotypic and multitypic response | eight months
  Monotypic: antibodies against one serotype Multitypic: antibodies against more than one serotype

CONTACTS AND LOCATIONS:
Locations (1):
- Mexican Society of Public Health, Mexico City, Mexico

REFERENCES:
- [Background] Organización Panamericana de la Salud. Dengue 2021 available at http://www.openepi.com/Menu/OE_Menu.htm
- [Background] Secretaria de Salud. Lineamientos para la vigilancia por laboratorio del dengue y otros arbovirus 2021. available at https://www.gob.mx/salud/documentos/lineamiento-estandarizado-para-la-vigilancia-epidemiologica-y-por-laboratorio-de-enfermedad-por-2019-ncov
- [Background] Centros para el Control y la Prevención de Enfermedades. Pruebas serológicas del virus del dengue 2020 [Available from: https://www.cdc.gov/dengue/es/healthcare-providers/testing/serologic-tests.html.
- [Background] Bhatt S, Gething PW, Brady OJ, Messina JP, Farlow AW, Moyes CL, Drake JM, Brownstein JS, Hoen AG, Sankoh O, Myers MF, George DB, Jaenisch T, Wint GR, Simmons CP, Scott TW, Farrar JJ, Hay SI. The global distribution and burden of dengue. Nature. 2013 Apr 25;496(7446):504-7. doi: 10.1038/nature12060. Epub 2013 Apr 7. PMID 23563266
- [Background] Organización Mundial de la Salud. Vacuna contra el dengue. Documento de posicion. Boletin Epidemiológico semanal 2018 36:457-76. available at https://www.who.int/immunization/policy/position_papers/PP_dengue_2018_SP.pdf?ua=1
- [Background] Katzelnick LC, Harris E; Participants in the Summit on Dengue Immune Correlates of Protection. Immune correlates of protection for dengue: State of the art and research agenda. Vaccine. 2017 Aug 24;35(36):4659-4669. doi: 10.1016/j.vaccine.2017.07.045. Epub 2017 Jul 28. PMID 28757058
- [Background] Martinez-Vega RA, Danis-Lozano R, Diaz-Quijano FA, Velasco-Hernandez J, Santos-Luna R, Roman-Perez S, Kuri-Morales P, Ramos-Castaneda J. Peridomestic Infection as a Determining Factor of Dengue Transmission. PLoS Negl Trop Dis. 2015 Dec 15;9(12):e0004296. doi: 10.1371/journal.pntd.0004296. eCollection 2015 Dec. PMID 26671573
- [Background] Amaya-Larios IY, Martinez-Vega RA, Mayer SV, Galeana-Hernandez M, Comas-Garcia A, Sepulveda-Salinas KJ, Falcon-Lezama JA, Vasilakis N, Ramos-Castaneda J. Seroprevalence of neutralizing antibodies against dengue virus in two localities in the state of Morelos, Mexico. Am J Trop Med Hyg. 2014 Nov;91(5):1057-65. doi: 10.4269/ajtmh.14-0145. Epub 2014 Oct 6. PMID 25294613
- [Background] World Health Organization. WHO Vaccine pipeline tracker 2020 [01/05/2021]. Available from: ttps://www.who.int/immunization/research/vaccine_pipeline_tracker_spreadsheet/en/.
- [Background] Hadinegoro SR, Arredondo-Garcia JL, Capeding MR, Deseda C, Chotpitayasunondh T, Dietze R, Muhammad Ismail HI, Reynales H, Limkittikul K, Rivera-Medina DM, Tran HN, Bouckenooghe A, Chansinghakul D, Cortes M, Fanouillere K, Forrat R, Frago C, Gailhardou S, Jackson N, Noriega F, Plennevaux E, Wartel TA, Zambrano B, Saville M; CYD-TDV Dengue Vaccine Working Group. Efficacy and Long-Term Safety of a Dengue Vaccine in Regions of Endemic Disease. N Engl J Med. 2015 Sep 24;373(13):1195-206. doi: 10.1056/NEJMoa1506223. Epub 2015 Jul 27. PMID 26214039
- [Background] Agocs MM, Serhan F, Yen C, Mwenda JM, de Oliveira LH, Teleb N, Wasley A, Wijesinghe PR, Fox K, Tate JE, Gentsch JR, Parashar UD, Kang G; Department of Immunization, Vaccines, and Biologicals, World Health Organization (WHO), Geneva, Switzerland; Centers for Disease Control and Prevention (CDC). WHO global rotavirus surveillance network: a strategic review of the first 5 years, 2008-2012. MMWR Morb Mortal Wkly Rep. 2014 Jul 25;63(29):634-7. PMID 25055187
- [Background] Biswal S, Borja-Tabora C, Martinez Vargas L, Velasquez H, Theresa Alera M, Sierra V, Johana Rodriguez-Arenales E, Yu D, Wickramasinghe VP, Duarte Moreira E Jr, Fernando AD, Gunasekera D, Kosalaraksa P, Espinoza F, Lopez-Medina E, Bravo L, Tuboi S, Hutagalung Y, Garbes P, Escudero I, Rauscher M, Bizjajeva S, LeFevre I, Borkowski A, Saez-Llorens X, Wallace D; TIDES study group. Efficacy of a tetravalent dengue vaccine in healthy children aged 4-16 years: a randomised, placebo-controlled, phase 3 trial. Lancet. 2020 May 2;395(10234):1423-1433. doi: 10.1016/S0140-6736(20)30414-1. Epub 2020 Mar 17. PMID 32197105
- [Background] Brunkard JM, Robles Lopez JL, Ramirez J, Cifuentes E, Rothenberg SJ, Hunsperger EA, Moore CG, Brussolo RM, Villarreal NA, Haddad BM. Dengue fever seroprevalence and risk factors, Texas-Mexico border, 2004. Emerg Infect Dis. 2007 Oct;13(10):1477-83. doi: 10.3201/eid1310.061586. PMID 18257990
- [Background] Navarrete-Espinosa J, Acevedo-Vales JA, Huerta-Hernandez E, Torres-Barranca J, Gavaldon-Rosas DG. [Prevalence of dengue and leptospira antibodies in the state of Veracruz, Mexico]. Salud Publica Mex. 2006 May-Jun;48(3):220-8. doi: 10.1590/s0036-36342006000300006. Spanish. PMID 16813130
- [Background] Amaya-Larios IY, Martinez-Vega RA, Diaz-Quijano FA, Sarti E, Puentes-Rosas E, Chihu L, Ramos-Castaneda J. Risk of dengue virus infection according to serostatus in individuals from dengue endemic areas of Mexico. Sci Rep. 2020 Nov 4;10(1):19017. doi: 10.1038/s41598-020-75891-z. PMID 33149151
- [Background] Amaya-Larios IY, Rojas-Russell M, Lopez-Cervantes M, Castro-Porras L, Castro-Borbonio MV, Sarti E, Puentes-Rosas E, Tirado-Gomez LL, Olaiz-Fernandez G, Ramos-Castaneda J. Seroprevalence of dengue in school children in Mexico ages 6-17 years, 2016. Trans R Soc Trop Med Hyg. 2018 May 1;112(5):223-229. doi: 10.1093/trstmh/try046. PMID 29917129
- [Background] Kaslow DC. Force of infection: a determinant of vaccine efficacy? NPJ Vaccines. 2021 Apr 12;6(1):51. doi: 10.1038/s41541-021-00316-5. PMID 33846340
- [Background] Gonzalez Morales NL, Nunez-Lopez M, Ramos-Castaneda J, Velasco-Hernandez JX. Transmission dynamics of two dengue serotypes with vaccination scenarios. Math Biosci. 2017 May;287:54-71. doi: 10.1016/j.mbs.2016.10.001. Epub 2016 Oct 20. PMID 27773682
- [Background] Schulte A, Weber I, Tiga-Loza DC, Amaya Larios IY, Shepard DS, Tschampl CA, Undurraga EA, Martinez-Vega RA, Fischer F, Chihu L, Ramos-Castaneda J. Health-Related Quality of Life after Dengue Fever, Morelos, Mexico, 2016-2017. Emerg Infect Dis. 2020 Apr;26(4):751-755. doi: 10.3201/eid2604.190729. PMID 32186487
- [Background] Pavia-Ruz N, Barrera-Fuentes GA, Villanueva-Jorge S, Che-Mendoza A, Campuzano-Rincon JC, Manrique-Saide P, Rojas DP, Vazquez-Prokopec GM, Halloran ME, Longini IM, Gomez-Dantes H. Dengue seroprevalence in a cohort of schoolchildren and their siblings in Yucatan, Mexico (2015-2016). PLoS Negl Trop Dis. 2018 Nov 21;12(11):e0006748. doi: 10.1371/journal.pntd.0006748. eCollection 2018 Nov. PMID 30462654